CLINICAL TRIAL: NCT05596019
Title: Effectiveness of Specific Neurodynamic Exercises Compared With Non-specific Exercises on Disability and Neck Pain in Women Older Than 65 Years
Brief Title: Specific Neurodynamic Exercises on Disability and Neck Pain in Old Women
Acronym: USNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Roberto Méndez Sánchez, Associate Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USalamancaNeckPain
Record Dates: First submitted 2022-10-19; First posted 2022-10-27 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Neck Pain
Keywords: exercise; neck pain; neurodynamic; elderly
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Longitudinal prospective, controlled, single-blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blind masking with blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neurodynamics specific exercise group (Experimental): The experimental group will perform a multimodal therapeutic physical exercise program. The components of balance, walking, cardiovascular endurance, strength and flexibility will be worked globally, in addition to including respiratory exercises.
  Specific neurodynamic exercises oriented to the treatment of the main nerves of the brachial plexus will be included as part of the exercise sessions. The specific neurodynamic program will consist of the following exercises:
  1. Opening of the cervical conjunction holes with cranio-cervical and cervical flexion movements, cervical lateroflexions and lateral vertebral sliding self-mobilizations.
  2. Opening of the thoracic passages of the brachial plexus with stretching of the scalene muscles, opening of the costoclavicular space and stretching of the pectoralis minor muscles.
  3. Specific exercises of neurodynamic sliding of the nerves of the upper limb: median, radial and ulnar nerves.
  Interventions: Procedure: specific neurodynamic exercises
- The nonspecific exercise group (Active Comparator): The nonspecific exercise group performed balance, cardiovascular endurance, stability, upper and lower limb strength, flexibility, and breathing exercises.
  Interventions: Procedure: multimodal exercise

INTERVENTIONS:
Procedure: specific neurodynamic exercises — Specific neurodynamic exercises in women older than 65 years with neck pain
  Arms: neurodynamics specific exercise group
Procedure: multimodal exercise — Multimodal and nonspecific exercises in women older than 65 years with neck pain
  Arms: The nonspecific exercise group

SUMMARY:
This is a randomized, parallel, double-blind clinical trial. The main objective is to compare the efficacy of multimodal exercise with specific neurodynamic exercises and multimodal exercise with non-specific exercises in disability and neck pain in women older than 65 years.

The intervention in both groups will be carried out for 4 weeks, with three weekly sessions. Two evaluations will be carried out, a pre-intervention evaluation and a post-intervention evaluation. We will assess neck pain, disability, upper limb strength, cervical mobility, cervical pressure pain thresholds, kinesiophobia and catastrophism.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 65 years.
* Neck pain

Exclusion Criteria:

* Tumors
* Pacemakers
* Fibrillations
* Cardiac pathology or uncontrolled hypertension
* History of severe trauma/recent cervical surgery
* Uncontrolled systemic and inflammatory pathologies
* Congenital collagen compromise
* Presence of difficulties in performing the Initial Evaluation tests
* Language barriers
* Pending litigation or legal claim

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-07-16 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity | four weeks.
  Numerical Pain Rating Scale (NPRS) will be used. It is a scale used to quantify the patient's pain level on an 11-point numerical scale 0-10 with 0 being "no pain" and 10 being the "worst possible pain."
Neck disability | four weeks
  The Neck Disability Index (NDI) will be used. It is a modification of the Oswestry Low Back Pain Disability Index. It is a scale used to measure disability associated with cervical pain due to acute or chronic conditions. He has 10 items: 7 related to activities of daily living, 2 related to pain and 1 related to concentration. The test can be interpreted with a maximum score of 50.

SECONDARY OUTCOMES:
Cervical range of motion | four weeks
  The Cervical Range of Motion (CROM) device (Performance Attainment Associates, USA) will be used to measure the cervical range of motion, including flexion, extension, lateral flexion and rotation.
Hand grip strength | four weeks
  The strength will be recorded with Jamar Plus: Digital dynamometer to assess grip strength.
upper limb strength | four weeks
  The strength in upper limb movements will be recorded with the device "wireless MicroFET 2": Hand-held dynamometer for force assessment.
Pressure pain threshold | four weeks
  Pressure algometry measurements will be performed with a digital algometer to assess pressure pain thresholds. (Algometer model: Pain Test™ FPIX 10).
Kinesiophobia | four weeks
  The Tampa Scale for kinesiophobia (TSK-13) will be used. It is a patient-reported outcome measure designed to help identify kinesiophobia. This version is a 13-item questionnaire aimed at the assessment of fear of movement/re-injury. Each item is provided with a 4-points Likert scale with scoring alternatives ranging from "strongly disagree" [0] to "strongly agree" [4] . This gives a possible total raw score range from 0 to 52.
Catastrophism | four weeks
  Pain Catastrophizing Scale (PCS) will be used. People are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Méndez-Sánchez, PhD, Principal Investigator — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Spain